CLINICAL TRIAL: NCT00346125
Title: An Evaluation of PET/CT Imaging as a Predictor of Disease Free Survival Following Neo-Adjuvant Chemotherapy for Soft Tissue Sarcoma
Brief Title: PET CT as Predictor of Response in Preoperative Chemotherapy for Soft Tissue Sarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2005LS080; UMN-0512M78446 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Sarcoma
Keywords: soft tissue sarcoma; Malignant fibrous histiocytoma; Liposarcoma; Fibrosarcoma; Leiomyosarcoma; Synovial sarcoma; Malignant peripheral nerve sheath tumor (MPNST); Epithelioid sarcoma
MeSH Terms: conditions — Sarcoma; Histiocytoma, Malignant Fibrous; Liposarcoma; Fibrosarcoma; Leiomyosarcoma; Sarcoma, Synovial; Neurofibrosarcoma | interventions — pegfilgrastim; Doxorubicin; Ifosfamide; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preferred Standard Regimen (Active Comparator): Subjects with soft tissue sarcoma who are receiving pegylated liposomal doxorubicin hydrochloride, Ifosfamide with mesna and pegfilgrastim - Repeat every 28 days for 4 cycles total
  Interventions: Biological: pegfilgrastim; Drug: ifosfamide; Drug: pegylated liposomal doxorubicin hydrochloride; Procedure: conventional surgery; Radiation: fludeoxyglucose F 18
- Alternative Treatment Regimen (Active Comparator): Subjects with soft tissue sarcoma who are receiving Doxorubicin hydrochloride, Ifosfamide with mesna and pegfilgrastim - Repeat every 28 days for 4 cycles total
  Interventions: Biological: pegfilgrastim; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Procedure: conventional surgery; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Biological: pegfilgrastim — will be given at 6 mg subcutaneously (SC) at the end of the mesna infusion
  Other Names: Neulasta(R)
Drug: doxorubicin hydrochloride — 65 mg/m^2 by continuous intravenous (IV) infusion over 7 days beginning on day 1
  Other Names: Doxorubicin; Adriamycin
  Arms: Alternative Treatment Regimen
Drug: ifosfamide — 9 g/m^2 by continuous intravenous (IV) infusion over 6 days beginning on day 1 with mesna 10.5 g/m^2 by continuous IV infusion over 7 days beginning on day 1
  Other Names: Mitoxana; Ifex
Drug: pegylated liposomal doxorubicin hydrochloride — 45 mg/m2 intravenous (IV) Day 1, repeat every 28 days.
  Other Names: doxorubicin-hydrochloride-liposome
  Arms: Preferred Standard Regimen
Procedure: conventional surgery — The surgical procedure will be decided by the treating physician and independent of study participation
Radiation: fludeoxyglucose F 18 — FDG is a radioactive sugar equal to a uniform whole-body exposure of approximately 1.5 rem for each scan. Post-operative radiation therapy may be given according to institutional guidelines in patients felt to have close surgical margins.
  Other Names: FDG

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography (PET) scan and computated tomography (CT) scan, may help doctors predict a patient's response to treatment and may help plan the best treatment. Drugs used in chemotherapy, such as doxorubicin and ifosfamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This clinical trial is studying how well PET scan combined with CT scan predicts response in patients undergoing chemotherapy and surgery for soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether measurements of fludeoxyglucose (FDG) positron emission tomography (PET)/CT imaging can accurately predict disease-free survival of patients with soft tissue sarcoma who are receiving neoadjuvant chemotherapy.

Secondary

* Correlate histological response to neoadjuvant chemotherapy for soft tissue sarcomas with FDG-PET/CT imaging findings.

Tertiary

* Determine the changes in FDG-PET/CT imaging over time as each course of chemotherapy is given.

OUTLINE: Patients receive 1 of 2 standard chemotherapy regimens:

* Preferred regimen: Patients receive pegylated doxorubicin HCl liposome IV on day 1, ifosfamide IV continuously on days 1-6, and pegfilgrastim subcutaneously (SC) on day 8. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Alternative regimen: Patients receive doxorubicin hydrochloride IV continuously on days 1-7. Patients also receive ifosfamide and pegfilgrastim as in the preferred regimen. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

All patients undergo a fludeoxyglucose positron emission tomography/CT scan at baseline, after course 1, and after completion of chemotherapy. Patients undergo surgery within 4-6 weeks after completion of chemotherapy.

After completion of study treatment and surgery, patients are followed every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 62 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, high grade, soft tissue sarcoma including

  * malignant fibrous histiocytoma,
  * liposarcoma,
  * fibrosarcoma,
  * leiomyosarcoma,
  * synovial carcinoma,
  * malignant peripheral nerve sheath tumor (MPNST),
  * epithelioid sarcoma, and
  * sarcomas-not otherwise specified.

NOTE: Ewings sarcoma, primitive neuroectodermal tumor, extraskeletal, osteosarcoma, extraskeletal chondrosarcoma, alveolar soft part sarcoma, rhabdomyosarcoma, carcinosarcoma, Kaposi's sarcoma, angiosarcoma, and mesothelioma patients are ineligible for this study.

* Measurable disease using traditional cross section measurements with the primary site's largest diameter > 5 centimeters by positron emission tomography/computated tomography (PET/CT), CT or magnetic resonance imaging (MRI) scan. Patients with either localized (primary or locally recurrent) or metastatic disease at presentation are eligible for study if they are to receive neoadjuvant treatment prior to excision of the primary (stage IIC, III, IVA, IVB.)
* Age ≥ 16 years, Karnofsky ≥ 70%
* Adequate organ function for receiving chemotherapy as determined by the treating physician.
* Women of childbearing potential and sexually active males are required to use an effective method of contraception (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the study.

Exclusion Criteria:

* Previous treatment with chemotherapy or radiation therapy
* Females known to be pregnant or breast-feeding are excluded because PET/CT scan in pregnant women is not FDA approved.
* Serious concomitant systemic disorders (eg, active infection) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study. Patients with PET-CT as an indicator of disease survival in soft tissue sarcoma untreated or symptomatic CNS metastases or uncontrolled diabetes will not be eligible.

Patient must give written informed consent indicating the investigational nature of the study and its potential risks.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-04-10 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | Baseline through Survival Event
  Compare changes in baseline and follow-up fludeoxyglucose (FDG) positron emission tomography (PET)/CT imaging with disease-free survival by peak SUV and max SUV calculations. Changes in baseline and follow-up PET/CT, based on max SUV calculations, will be compared with disease free survival. Disease free survival will be measured in months from the time of study enrollment until the time that disease recurrence/relapse/progression is recorded.

SECONDARY OUTCOMES:
Correlate histologic response with FDG-PET/CT imaging | At end of each cycle
  The overall histologic response will be defined as:
  % histologic response = 100 - % viable tumor in the central slice as assessed histologically It should be noted that the % histologic response is different from % tumor necrosis as it includes an assessment of the % tumor necrosis along with the degenerative changes
Compare changes in FDG-PET/CT imaging with disease-free survival by max SUV calculations | Baseline Compared to 1 Cycle and Baseline to After Chemotherapy
  Changes in PET/CT from baseline will be compared to PET/CT done after one cycle and after completion of chemotherapy treatment before surgical excision using max SUV calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Cheng, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Derived] O'Donnell PW, Manivel JC, Cheng EY, Clohisy DR. Chemotherapy influences the pseudocapsule composition in soft tissue sarcomas. Clin Orthop Relat Res. 2014 Mar;472(3):849-55. doi: 10.1007/s11999-013-3022-7. PMID 23640206